CLINICAL TRIAL: NCT05427240
Title: A Randomized Hybrid Type I Effectiveness-Implementation Study of an eHealth Delivery Alternative for Cancer Genetic Testing for Hereditary Cancer
Brief Title: eHealth Delivery Alternative for Cancer Genetic Testing for Hereditary Cancer
Acronym: eReach2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Fox Chase Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 13021; 850242 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2022-06-07; First posted 2022-06-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ARM A (Experimental): Visit 1/Pre-Test Session - Standard-of-Care Pre-Test Counseling with a genetic counselor.
  Visit 2/Disclosure Session - Standard-of-Care Post-Test Counseling with a genetic counselor.
  Interventions: Other: Standard of Care
- ARM B (Experimental): Visit 1/Pre-Test Session - Standard-of-Care Pre-Test Counseling with a genetic counselor.
  Visit 2/Disclosure Session - Self-directed web-based eHealth result disclosure intervention.
  Interventions: Other: Pre-Test Intervention; Other: Standard of Care
- ARM C (Experimental): Visit 1/Pre-Test Session - Self-directed web-based eHealth pre-test session intervention.
  Visit 2/Disclosure Session - Standard-of-Care Post-Test Counseling with a genetic counselor.
  Interventions: Other: Standard of Care; Other: Post-Test Intervention
- ARM D (Experimental): Visit 1/Pre-Test Session - Self-directed web-based eHealth pre-test session intervention.
  Visit 2/Disclosure Session - Self-directed web-based eHealth result disclosure intervention.
  Interventions: Other: Pre-Test Intervention; Other: Post-Test Intervention

INTERVENTIONS:
Other: Pre-Test Intervention — Secure and accessible by private code only, the web-based intervention will provide users with a the results of their clinical genetic testing results and a detailed summary of what those results mean. Additionally, an individualized summary will also be included.
  Arms: ARM B; ARM D
Other: Standard of Care — Standard of Care with a Genetic Counselor by Remote Services
  Arms: ARM A; ARM B; ARM C
Other: Post-Test Intervention — Secure and accessible by private code only, the web-based intervention will provide users with a the results of their clinical genetic testing results and a detailed summary of what those results mean. Additionally, an individualized summary will also be included.
  Arms: ARM C; ARM D

SUMMARY:
This randomized non-inferiority study will use a 2x2 design where traditional standard-of-care pre-test (visit 1) and post-test (visit 2: disclosure) counseling delivered by a genetic counselor are replaced with a self-directed web-based eHealth intervention to provide critical data to inform optimal ways to deliver clinical genetic testing in eligible individuals, while maintaining quality of care and favorable cognitive, affective and behavioral outcomes.

DETAILED DESCRIPTION:
Germline cancer genetic testing has become a standard evidence-based practice, with established risk reduction and cancer screening guidelines for genetic carriers. Access to genetic specialists is limited in many areas in the US, and the traditional medical delivery model of pre- and post-test counseling with a genetic professional will not support the rising indications for genetic testing. Recent data from the National Health Interview Survey found that <20% of eligible patients with a personal or family history of breast or ovarian cancer underwent genetic testing. Thus, there is an urgent need to consider alternative delivery models to increase access and uptake of genetic testing, while maintaining adequate patient cognitive, affective and behavioral outcomes.

This study aims to evaluate the effectiveness of offering web-based eHealth delivery alternatives of pre/post-test genetic counseling to provide equal or improved timely uptake of genetic services and testing, and short-term cognitive (e.g. understanding), affective (e.g. distress and uncertainty) and behavioral (risk reducing and screening behaviors and communication to providers and relatives) outcomes in patients with barriers to genetic testing as compared to the traditional two-visit delivery model with a genetic counselor.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Speak and understand English
* Male or Female
* No prior germline genetic testing
* Meet current National Comprehensive Cancer Network (NCCN) guidelines for germline genetic testing

Exclusion Criteria:

-Communication difficulties such as:

* Uncorrected or uncompensated hearing and/or vision impairment
* Uncorrected or uncompensated speech defects
* Uncontrolled psychiatric/mental condition or severe physical, neurological or cognitive deficits rendering individual unable to understand study goals and tasks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2025-12-24 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The KnowGene Scale | Through study completion, an average of 1 year
  Change in Knowledge - Score Range = 0-16, Higher score = Better outcome
Patient Reported Outcome Measurement Information System (PROMIS) | Through study completion, an average of 1 year
  Change in General Anxiety - Score Range = 4-20, Lower score = Better outcome
Uptake of Genetic Services | Through study completion, an average of 1 year
  Testing uptake per arm - Yes/No

SECONDARY OUTCOMES:
Patient Reported Outcome Measurement Information System (PROMIS) | Through study completion, an average of 1 year
  Change in General Depression - Score Range = 4-20, Lower score = Better outcome
Impact of Events Scale (IES) | Through study completion, an average of 1 year
  Change in Cancer Specific Distress - Score Range = 0-40, Lower score = Better outcome
Multi-dimensional Impact of Cancer Risk Assessment Questionnaire (MICRA) | Through study completion, an average of 1 year
  Change in Uncertainty - Score Range = 0-85, Lower score = Better outcome
Satisfaction with genetic services | Through study completion, an average of 1 year
  Differences in satisfaction by Arm - Score Range = 14-70, Higher score = Better outcome
Decisional Regret Scale | Through study completion, an average of 1 year
  Differences in decisional regret by Arm - Score Range = 5-25, Lower score = Better outcome
Provider Time | Through study completion, an average of 1 year
  Time (minutes) provider spends per patient

CONTACTS AND LOCATIONS:
Overall Officials: Angela R Bradbury, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mastaglio E, Egleston B, Lee KT, Fetzer D, Brown S, Domchek SM, Fleisher L, Wen KY, Wagner L, Roberts JS, Cacioppo C, Christiansen J, Howe S, Wood EM, Weinberg M, Karpink K, Selmani E, Feng J, John S, Schweickert K, McLeod B, Bradbury AR. A Randomized Hybrid Type I Effectiveness-Implementation Study of an eHealth Delivery Alternative for Cancer Genetic Testing for Hereditary Cancer (eREACH2): study protocol. medRxiv [Preprint]. 2025 Nov 22:2025.11.19.25340515. doi: 10.1101/2025.11.19.25340515. PMID 41332807